CLINICAL TRIAL: NCT05757778
Title: A Single-Blind, Split-Chest, Single-Center Study of the Effects of Breast Neurotization in Implant Based Breast Reconstruction
Brief Title: Split Chest Breast Neurotization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-01026
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Implant; Complications

STUDY DESIGN:
Who Masked: Participant
Masking Description: Within patients, treatment with neurotization to one breast will be randomly assigned intra-operatively. Patients will remain blinded from intraoperative details until the completion of the study. Patients will consent to remain blinded to the operative and postoperative reports until completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurotized Breast (Experimental): For patients undergoing bilateral implant-based breast reconstruction following nipple-sparing mastectomy, one breast will be neurotized by connecting the lateral intercostal nerve to the nipple with interposing standard nerve grafting techniques. The neurotized breast will serve as the "experimental" breast. The other breast will not receive any breast neurotizing procedure.
  Interventions: Procedure: Sensory Nerve Coaptation
- Non-Neurotized Breast (No Intervention): For patients undergoing bilateral implant-based breast reconstruction following nipple-sparing mastectomy, one breast will not receive any breast neurotizing procedure. The non-neurotized breast will serve as the "control" breast.

INTERVENTIONS:
Procedure: Sensory Nerve Coaptation — Nerve reconstruction will employ an off-the-shelf nerve graft coapted to the donor anterior intercostal nerve branch laterally and medially at the underside of the nipple. The anterior intercostal nerve branch and nerve graft coaptation will be performed in a standard fashion with a 1 mm gap between the ends of the graft and the donor nerve. Medially, the nerve graft will be inset into the underside of the preserved nipple-areola complex using 8-0 or 9-0 epineural stitches from the nerve allograft. All nerve coaptations will be performed under loupe magnification as is standardly performed.
  Arms: Neurotized Breast

SUMMARY:
Several members of the scientific community have suggested that breast neurotization can help return nipple sensation to patients undergoing implant-based breast reconstruction. There has been no randomized controlled study assessing the validity of these claims. The goal of this study is to evaluate if performing breast neurotization can help restore or improve return of nipple sensation to patients undergoing implant-based breast reconstruction. This will be a single-blinded, randomized controlled trial where patients undergoing bilateral reconstruction will serve as their own controls by receiving an intervention on one breast but not the other breast.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing bilateral nipple-sparing mastectomy (prophylactic or therapeutic) at a single institution
* Women receiving implant-based reconstruction (either direct to implant or tissue expander-based implant reconstruction of any size)
* Age 18 or older

Exclusion Criteria:

* Women with history of prior breast surgery given concern for potentially damaged nerves by prior intervention that could impact the procedure and results. Procedures include but are not limited to: prior breast reduction, prior breast augmentation, prior lumpectomy
* Pre-operative radiation or anticipated post-operative radiation
* Body Mass Index (BMI) > 30 kg/m2 or patients with macromastia (larger breasts) as these patients frequently require larger implants that will not accommodate the longest nerve graft available (70 mm)
* Current tobacco or nicotine use
* History of diabetes mellites with a HgbA1c > 7% due to lower rates of wound healing
* History of auto-immune disease
* History of allergy, sensitivity, or intolerance to porcine-derived materials
* Intraoperatively, patients may have to be excluded if during the mastectomy the lateral nerve targets were severely damaged or removed as part of the mastectomy. While these patients will be excluded from the formal analysis, the investigators will continue to follow them as a subgroup for analysis and comparison.
* Men as they infrequently receive bilateral mastectomies due to breast cancer. Male breast cancer is <1% of all breast malignancies.
* Pregnancy as determined by urine pregnancy test on day of surgery

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Semmes-Weinstein Monofilament Testing (SWMT) Score in the Nipple (Area 9) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Nipple (Area 9) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.

SECONDARY OUTCOMES:
SWMT Score in the Mastectomy Superior (Area 1) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Superior (Area 1) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Lateral (Area 2) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Lateral (Area 2) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Inferior (Area 3) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Inferior (Area 3) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Medial (Area 4) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Mastectomy Medial (Area 4) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Superior (Area 5) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Superior (Area 5) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Lateral (Area 6) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Lateral (Area 6) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Inferior (Area 7) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Inferior (Area 7) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Medial (Area 8) | Month 12 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.
SWMT Score in the Flap Medial (Area 8) | Month 24 Post-Surgery
  SWMT will be used for assessment of breast sensation by applying the monofilament to a given anatomic region. Based on the monofilament size, a score of 0-6 is assigned. Scores are classified as follows: 6 = normal; 5 = diminished light touch; 4 = diminished protective sensation; 3 = loss of protective sensation; 2 = Loss of protective/sensation; 1 = Deep pressure sensation only; and 0 = Loss of sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Mihye Choi, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Thomas.Calahan@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.